CLINICAL TRIAL: NCT05620823
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled, Efficacy and Safety Study of Povorcitinib (INCB054707) in Participants With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study to Evaluate the Efficacy and Safety of Povorcitinib (INCB054707) in Participants With Moderate to Severe Hidradenitis Suppurativa
Acronym: STOP-HS1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB 54707-301; 2022-501752-29-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2022-11-10; First posted 2022-11-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Hidradenitis Suppurativa; Hidradenitis; Acne inversa; HS; INCB054707; Povorcitinib
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1:1 to Povorcitinib Dose A, Povorcitinib Dose B, or placebo once a day (QD); participants who complete the placebo controlled (PC) 12-week period may continue to a 42-week extension(EXT) period with Povorcitinib (Dose A or Dose B) QD.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Povorcitinib Dose A (Experimental): Participants will receive Povorcitinib Dose A for 54 weeks.
  Interventions: Drug: Povorcitinib
- Povorcitinib Dose B (Experimental): Participants will receive Povorcitinib Dose B for 54 weeks.
  Interventions: Drug: Povorcitinib
- Placebo (Placebo Comparator): Participants will receive Placebo for 12 weeks, followed by Povorcitinib (Dose A or Dose B) for 42 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Povorcitinib — Oral; Tablet
  Other Names: INCB054707
  Arms: Povorcitinib Dose A; Povorcitinib Dose B
Drug: Placebo — Oral; Tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Povorcitinib (INCB054707) in participants with moderate to severe Hidradenitis Suppurativa (HS) over a 12-week placebo controlled period, followed by a 42-week extension period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe HS for at least 3 months prior to the screening visit.
* Total abscess and inflammatory nodule count of at least 5 at both the screening and baseline visits
* HS lesions in at least 2 distinct anatomical areas (examples include but are not limited to left and right axilla or left and right inguinocrural fold), 1 of which must be at least Hurley Stage II or Hurley Stage III, at both the screening and baseline visits
* Documented history of inadequate response to at least a 3-month course of at least 1 conventional systemic therapy (oral antibiotic or biologic drug) for HS (or demonstrated intolerance to, or have a contraindication to, a conventional systemic therapy for treatment of their HS).
* Agreement to NOT use topical and systemic antibiotics for treatment of HS during the placebo-controlled period.
* Agreement to NOT use a diluted bleach bath or topical antiseptic washes containing chlorhexidine gluconate or benzoyl peroxide on the areas affected by HS lesions during the placebo-controlled period. Note: Over-the-counter soap and water is allowed.
* Agreement to use contraception
* Willing and able to comply with the study protocol and procedures.
* Further inclusion criteria apply.

Exclusion Criteria:

* Presence of > 20 draining tunnels (fistulas) at either the screening or baseline visit.
* Women who are pregnant (or who are considering pregnancy) or breastfeeding.
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction, Q-wave interval abnormalities, current or history of certain infections, cancer, lymphoproliferative disorders and other medical conditions at the discretion of the investigator.
* Laboratory values outside of the protocol-defined ranges.
* Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who achieve Hidradenitis Suppurativa Clinical Response (HiSCR) | Week 12
  HiSCR is defined as at least a 50% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining tunnel count.

SECONDARY OUTCOMES:
Proportion of participants who achieve Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) | Week 12
  HiSCR75 is defined as at least a 75% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining tunnel count.
Proportion of participants with flare | 12 weeks
  Participants who experience at least 1 flare over 12 weeks; flare is defined as at least a 25% increase in the total abscess and inflammatory nodule count with a minimum increase of 2 relative to baseline.
Proportion of participants with a ≥ 3-point decrease in Skin Pain Numeric Rating Scale (NRS) score among participants with baseline Skin Pain NRS score ≥ 3. | Week 12
  Participants with a Skin Pain score of at least 3 at baseline and who experience at least a 3-point decrease in Skin Pain score at Week 12, relative to baseline. Skin Pain is an 11 point NRS, ranging from 0 (no skin pain) to 10 (worst skin pain).
Proportion of participants who achieve Skin Pain NRS30 among participants with baseline Skin Pain NRS score ≥ 3. | Week 12
  Participants with a Skin Pain score of at least 3 at baseline and who achieve at Week 12 Skin Pain NRS30, defined as at least a 30% reduction and at least 1-unit reduction from baseline in the Skin Pain NRS.
Proportion of participants with a ≥ 4-point increase from baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT F) score | Week 12
  Participants with a baseline FACIT-F score ≤ 48 and who experience at least a 4-point increase in FACIT-F score at Week 12, relative to baseline. The FACIT-F scale is a 13-item questionnaire that assesses self reported fatigue and its impact upon daily activities and function over the past 7 days, with scores ranging from 0 (worst fatigue) to 52 (no fatigue).
Mean change from baseline in Dermatology Life Quality Index (DLQI) score at each visit | 54 weeks
  The DLQI is a skin disease specific questionnaire aimed at the evaluation of how symptoms and treatment affect participants' health-related quality of life (QoL). The DLQI total score ranges from 0 to 30, with higher scores indicating lower skin health related QoL.
Mean change from baseline in abscess count at each visit. | 54 weeks
  Defined as mean change of Abscess count relative to baseline.
Percentage change from baseline in abscess count at every visit | 54 weeks
  Percent change from baseline in number of abscess(es)
Mean change from baseline in inflammatory nodule count at each visit | 54 weeks
  Defined as mean change of inflammatory nodule count relative to baseline.
Percentage change from baseline in inflammatory nodule count at each visit. | 54 weeks
  Defined as percent change from baseline in number of inflammatory nodule(s)
Mean change from baseline in draining tunnel count at each visit. | 54 weeks
  Defined as mean change of draining tunnel count relative to baseline.
Percentage change from baseline in draining tunnel count at each visit. | 54 weeks
  Defined as percent change from baseline in number of draining tunnel(s)
Extension Period: Proportion of participants who achieve HiSCR | Week 24
  HiSCR is defined as at least a 50% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining tunnel count.
Extension Period: Proportion of participants who achieve HiSCR75 | Week 24
  HiSCR75 is defined as at least a 75% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining tunnel count.
Extension Period: Proportion of participants with flare | From Week 12 through Week 24
  Participants who experience at least 1 flare over the period under assessment; flare is defined as at least a 25% increase in the total abscess and inflammatory nodule count with a minimum increase of 2 relative to baseline.
Extension Period: Proportion of participants who achieved Skin Pain NRS30 among participants with baseline Skin Pain NRS score ≥ 3 | Week 24
  Skin Pain NRS30 defined as at least a 30% reduction and at least 1-unit reduction from baseline in the Skin Pain NRS.
Extension Period: Proportion of participants who achieve HiSCR | Week 54
  HiSCR is defined as at least a 50% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining tunnel count
Extension Period: Proportion of participants who achieve HiSCR75 | Week 54
  HiSCR75 is defined as at least a 75% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining tunnel count.
Extension Period : Proportion of participants with flare | From Week 12 through Week 54
  Participants who experience at least 1 flare over the period under assessment; flare is defined as at least a 25% increase in the total abscess and inflammatory nodule count with a minimum increase of 2 relative to baseline.
Extension Period: Proportion of participants who achieved Skin Pain NRS30 among participants with baseline Skin Pain NRS score ≥ 3. | Week 54
  Participants with a Skin Pain score of at least 3 at baseline and who achieve at Week 24 Skin Pain NRS30, defined as at least a 30% reduction and at least 1-unit reduction from baseline in the Skin Pain NRS.
Extension Period:Proportion of participants who achieve maintenance of HiSCR or greater response at each visit | From Week 12 through Week 54
  Maintenance of response defined as participants who achieve HiSCR at Week 12 and maintain it or achieve greater response at each visit during the EXT period.
Extension Period : Proportion of participants who achieve maintenance of HiSCR75 or greater response at each visit | From Week 12 through Week 54
  Maintenance of response defined as participants who achieve HiSCR75 at Week 12 and maintain it or achieve greater response at each visit during the EXT period.

CONTACTS AND LOCATIONS:
Locations (104):
- United States (37):
  - Investigative Site US303, Phoenix, Arizona
  - Investigative Site US335, Arkansas City, Arkansas
  - Investigative Site US307, Fort Smith, Arkansas
  - Investigative Site US315, Laguna Niguel, California
  - Investigative Site US326, Los Angeles, California
  - Investigative Site US323, San Francisco, California
  - Investigative Site US306, Boca Raton, Florida
  - Investigative Site US320, Boca Raton, Florida
  - Investigative Site US317, Hialeah, Florida
  - Investigative Site US338, Margate, Florida
  - Investigative Site US321, North Miami Beach, Florida
  - Investigative Site US316, Orlando, Florida
  - Investigative Site US328, Tampa, Florida
  - Investigative Site US336, Tampa, Florida
  - Investigative Site US311, Marietta, Georgia
  - Investigative Site US327, Chicago, Illinois
  - Investigative Site US319, Skokie, Illinois
  - Investigative Site US337, Indianapolis, Indiana
  - Investigative Site US341, Bowling Green, Kentucky
  - Investigative Site US334, Metairie, Louisiana
  - Investigative Site US333, Baltimore, Maryland
  - Investigative Site US325, Columbia, Maryland
  - Investigative Site US318, Beverly, Massachusetts
  - Investigative Site US304, Boston, Massachusetts
  - Investigative Site US310, Brighton, Massachusetts
  - Investigative Site US302, St Louis, Missouri
  - Investigative Site US331, Albuquerque, New Mexico
  - Investigative Site US324, Kew Gardens, New York
  - Investigative Site US339, Bexley, Ohio
  - Investigative Site US330, Boardman, Ohio
  - Investigative Site US314, Cincinnati, Ohio
  - Investigative Site US312, Cleveland, Ohio
  - Investigative Site US301, Portland, Oregon
  - Investigative Site US340, Bellaire, Texas
  - Investigative Site US300, Plano, Texas
  - Investigative Site US313, Norfolk, Virginia
  - Investigative Site US308, Spokane, Washington
- Austria (7):
  - Investigative Site AT304, Graz
  - Investigative Site 00A, Innsbruck
  - Investigative Site AT306, Innsbruck
  - Investigative Site AT302, Linz
  - Investigative Site AT305, Vienna
  - Investigative Site AT301, Vienna
  - Investigative Site AT300, Vienna
- Belgium (7):
  - Investigative Site BE300, Brussels
  - Investigative Site BE304, Brussels
  - Investigative Site BE301, Ghent
  - Investigative Site BE306, Ghent
  - Investigative Site BE305, Leuven
  - Investigative Site BE302, Liège
  - Investigative Site BE303, Namur
- Canada (8):
  - Investigative Site CA301, Winnipeg, Manitoba
  - Investigative Site CA304, Barrie, Ontario
  - Investigative Site CA308, Hamilton, Ontario
  - Investigative Site CA303, London, Ontario
  - Investigative Site CA302, Peterborough, Ontario
  - Investigative Site CA306, Laval, Quebec
  - Investigative Site CA307, Montreal, Quebec
  - Investigative Site CA309, Québec, Quebec
- Czechia (2):
  - Investigative Site CZ301, Ostrava - Poruba
  - Investigative Site CZ300, Prague
- France (8):
  - Investigative Site FR305, Bordeaux
  - Investigative Site FR303, Brest
  - Investigative Site FR307, Le Mans
  - Investigative Site FR304, Marseille
  - Investigative Site FR302, Nantes
  - Investigative Site FR300, Paris
  - Investigative Site FR301, Saint-Priest-en-Jarez
  - Investigative Site FR306, Toulouse
- Germany (8):
  - Investigative Site DE305, Darmstadt
  - Investigative Site DE302, Dresden
  - Investigative Site DE306, Düsseldorf
  - Investigative Site DE301, Frankfurt am Main
  - Investigative Site DE303, Hamburg
  - Investigative Site DE300, Hanover
  - Investigative Site DE304, Langenau
  - Investigative Site DE307, Memmingen
- Greece (4):
  - Investigative Site GR300, Athens
  - Investigative Site GR303, Athens
  - Investigative Site GR301, Thessaloniki
  - Investigative Site GR302, Thessaloniki
- Japan (10):
  - Investigative Site JP304, Itabashi-ku
  - Investigative Site JP305, Kurume-shi
  - Investigative Site JP300, Kyoto
  - Investigative Site JP301, Nakagami-gun
  - Investigative Site JP303, Niigata
  - Investigative Site JP307, Nishinomiya-shi
  - Investigative Site JP308, Sapporo
  - Investigative Site JP302, Sendai
  - Investigative Site JP309, Shinjuku-ku
  - Investigative Site JP306, Tsukuba
- Netherlands (3):
  - Investigative Site NL302, Breda
  - Investigative Site NL303, Groningen
  - Investigative Site NL301, Rotterdam
- Poland (4):
  - Investigative Site PL304, Ostrowiec
  - Investigative Site PL303, Poznan
  - Investigative Site PL301, Wroclaw
  - Investigative Site PL302, Wroclaw
- Spain (6):
  - Investigative Site ES302, Badalona
  - Investigative Site ES303, Barcelona
  - Investigative Site ES301, Granada
  - Investigative Site ES305, Madrid
  - Investigative Site ES300, Pontevedra
  - Investigative Site ES304, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Study to Evaluate the Efficacy and Safety of Povorcitinib (INCB054707) in Participants With Moderate to Severe Hidradenitis Suppurativa — https://incyteclinicaltrials.com/studies/incb-54707-301